CLINICAL TRIAL: NCT03862885
Title: Early Access Program (EAP) for Avapritinib in Patients With Locally Advanced Unresectable or Metastatic Gastrointestinal Stromal Tumor (GIST)
Brief Title: Early Access Program (EAP) for Avapritinib in Patients With Locally Advanced Unresectable or Metastatic GIST
Status: Approved for marketing | Type: Expanded Access
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BLU-285-EAP-01
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: GIST
MeSH Terms: interventions — avapritinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Avapritinib — Avapritinib will be administered orally (PO) at a dose of 300 mg once daily (QD) in continuous 28-day cycles.
  Other Names: BLU-285

SUMMARY:
This is a US, multicenter, open-label expanded access program to provide access to avapritinib until such time that avapritinib becomes available through other mechanisms or the Sponsor chooses to discontinue the program.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 16 years of age.
2. Diagnosis of unresectable or metastatic GIST
3. The patient is not eligible for an ongoing study of avapritinib or cannot access an ongoing study of avapritinib.
4. Patient has received 3 or more TKI therapies including imatinib, or the patient has GIST that carries a mutation in exon 18 of the PDGFRA gene (such as D842V).
5. The patient has adequate vital organ function, including heart, lungs, liver, kidneys, bone marrow and endocrine, and is expected to tolerate therapy with a TKI.
6. Patient or legal guardian, if permitted by local regulatory authorities, provides informed consent.

Exclusion Criteria:

1. Patients who have poor organ function as defined by one or more of the following laboratory parameters;

   1. Total bilirubin > 2 × ULN; or > 3 × ULN in the presence of Gilbert's Disease;
   2. Platelet count < 75 × 10^9/L.
2. Patient requires therapy with a concomitant medication that is a strong inhibitor or strong inducer of cytochrome P450 (CYP) 3A4
3. Patient has had a major surgical procedure (minor surgical procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures) within 14 days of the first dose of avapritinib.
4. Patient has a history of a cerebrovascular accident or transient ischemic attacks within 1 year prior to the first dose of program drug.
5. Patient has a known risk of intracranial bleeding, such as a brain aneurysm or history of subdural or subarachnoid bleeding.
6. Women who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of randomization and for at least 30 days after the last dose of avapritinib. Men who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of first dose and for at least 90 days after the last dose of avapritinib.
7. Women who are pregnant, as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy, obtained within 7 days before the randomization. Females with β-hCG values that are within the range for pregnancy but are not pregnant (false-positives) may be enrolled with written consent of the Sponsor, after pregnancy has been ruled out. Females of non- childbearing potential (postmenopausal for more than 1 year; bilateral tubal ligation; bilateral oophorectomy; hysterectomy) do not require a serum β-hCG test.
8. Women who are breast feeding.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult